CLINICAL TRIAL: NCT02969512
Title: Feasibility of the Hip Instructional Prehabilitation Program for Enhanced Recovery (HIPPER) Intervention Protocol: An eHealth Approach for Pre-surgical Hip Replacement Education
Brief Title: Feasibility of the Hip Instructional Prehabilitation Program for Enhanced Recovery (HIPPER)
Acronym: HIPPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, William C. Miller, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H16-02553
Record Dates: First submitted 2016-11-09; First posted 2016-11-21 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Hip Osteoarthritis
Keywords: Patient education; Advanced hip osteoarthritis; Online education; Computer-assisted instruction; e-learning; Older adult
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIPPER (Experimental): The HIPPER group will receive 12 interactive online modules (~20 minutes each). HIPPER participants will receive email or phone contact (participant preference) to provide them with website portal access consisting of the web address, and simple instructions to access the website using personalized encrypted login information to the site.
  Interventions: Other: HIPPER
- OASIS Online Educational Webinars (Active Comparator): To provide a comparable level of education, participants in the Online Education group will receive 2 hours of OASIS online educational webinars as per current practice.
  Interventions: Other: OASIS Online Educational Webinars

INTERVENTIONS:
Other: HIPPER — Participants can complete the online educational modules at home or another location with internet access. The total time to complete all of the modules is about 2 hours and 30 minutes.
  Other Names: Behavioral: Online prehab education
  Arms: HIPPER
Other: OASIS Online Educational Webinars — 2-hour online educational large group sessions
  Other Names: Behavioral: large group education sessions
  Arms: OASIS Online Educational Webinars

SUMMARY:
Osteoarthritis (OA), leading to hip replacement, is a leading contributor to global mobility impairment. Given the boom in the older demographic it is not surprising that there is an 11% increased demand for replacement every 5 years in Canada. Health promotion interventions, such as prehabilitation, defined as pre-surgical education, are vital to optimizing surgical outcomes, reducing hospitalization costs, accelerating rehabilitation, and reducing patient discomfort and pre-operative anxiety. HIPPER is a 2-year randomized controlled trial (RCT) that will assess feasibility indicators and clinical outcomes of online prehab education modules compared to online educational webinars. The feasibility indicators (process, resource, management, and treatment issues) and clinical outcomes (physical function, anxiety, depression, pain, daily activities, self-efficacy, and health related quality of life) will be assessed among Vancouver-dwelling older adults aged > 50 years, with advanced hip osteoarthritis. The findings will lead to the refinement of the design protocol in order to evaluate a contemporary, standardized, and geographically accessible prehab education program in a large multi-site RCT.

DETAILED DESCRIPTION:
This feasibility study will use a single-site, parallel group evaluator blind RCT. Subjects (N=40) will be randomly assigned to the experimental (HIPPER n=20) or control (n=20) groups.The experimental group will receive the interactive online HIPPER intervention consisting of 12 modules (~20 mins/module). The control group is usual practice consisting of a 2 hr online large group educational webinar. Feasibility indicators (i.e. recruitment and retention; subject burden; safety; intervention administration/adherence; perceived benefit) will be evaluated as binary outcomes against pre-set parameters reflecting viability for a multi-site large-scale RCT. The primary clinical outcome of interest when assessing effect size for the eventual RCT is the Hospital Anxiety and Depression Scale-Anxiety. Secondary clinical outcomes include measures of pain, function, daily activities, self-efficacy, equipment checklist, system usability scale, environmental setup, physical activity, and health related quality of life.

Upon successful screening/enrollment and baseline data collection (T1) the Study Coordinator will contact the statistician by telephone or email and obtain group assignment within 48 hours. Subjects will be randomized using a 1:1 allocation ratio between groups. A central computerized randomization process will be designed by the statistician, with an undisclosed block size. To address bias, subjects will be instructed not to discuss their program and Testers will reinforce this point at each session. T1 data will be collected at our clinic while the follow up data collected 7-10 days prior to surgery (T2), and 30 days post-surgery (T3).

The findings from the study will be summarized and mailed to each participant upon study completion. HIPPER and control group assessments will be held at GF Strong Rehabilitation Centre and at subject's homes.

The outcome will lead to the refinement of the design protocol in order to robustly evaluate a contemporary, standardized, and geographically accessible prehabilitation education program. Ultimately, HIPPER may be found to have significant individual and social (health system level) benefits.

ELIGIBILITY:
Inclusion Criteria:

Community-dwelling participants with advanced hip OA will be included if they:

* are living in the greater Vancouver region;
* are aged 50 years or older;
* are scheduled to have a single THR in 12 weeks or later;
* have access to the internet

Exclusion Criteria:

* cannot communicate and complete questionnaires in English;
* anticipate a health condition or procedure that contraindicates their THR surgery;
* are actively receiving physical therapy for their hip symptoms;
* have had a previous THR.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Change in Primary Clinical Outcomes Scale | Baseline,7-10 days before surgery, Post Intervention (30 days after surgery).
  Hospital Anxiety and Depression Scale (HADS-A): The HADS-A is a validated 7-item tool that includes tension, worry and fear and has respondents indicate how they currently feel on each item.

SECONDARY OUTCOMES:
30-second Chair-Stand Test | Baseline,7-10 days before surgery.
  Functional lower limb strength and dynamic balance will be assessed by having subjects perform repeated sit-to-stands using a standard 43-46 cm straight back chair with no arm rests.
Change in Physical Activity Scale for the Elderly (PASE) | Baseline,7-10 days before surgery, Post Intervention (30 days after surgery).
  Patients are less physically active prior to THR and show minimal improvements in activity levels post-operatively. PASE is 12-item tool developed for older adults to assess home, occupational and recreational activities in the previous 7 days.
Change in Self-Efficacy for Rehabilitation Outcome Scale (SER) | Baseline,7-10 days before surgery, Post Intervention (30 days after surgery).
  The SER is a 12-item questionnaire that asks patients to rate their confidence on an 11-point Likert scale and generates 2 subscale scores: self-efficacy for rehabilitation therapy exercises and self-efficacy for overcoming barriers.
Equipment Checklist | Baseline,7-10 days before surgery, Post Intervention (30 days after surgery).
  It is recommended that patients acquire equipment and mobility aids prior to THR to ensure their safety, carry out daily living activities and adhere to surgical precautions post-operatively. A comprehensive checklist of recommended equipment will be created based on current guidelines, clinical recommendations and our Patient Partners' input.
EuroQol-5 Dimension, 5 level | Baseline,7-10 days before surgery, Post Intervention (30 days after surgery).
  Health-related quality of life is a core outcome for hip OA and the EQ-5D a suggested measure. The EQ-5D is a brief questionnaire that assesses 5 health status domains, reflected in a single-score, and overall health state using a visual analogue scale.
System Usability Scale | 7-10 days before surgery, Post Intervention (30 days after surgery)
  System Usability Scale consists of a 10 item questionnaire with five response options for respondents; from "Strongly agree" to "Strongly disagree". Originally created by John Brooke in 1986, it allows to evaluate a wide variety of products and services, including hardware, software, mobile devices, websites and applications. Some example items are "I think that I would like to use this system frequently." and "I needed to learn a lot of things before I could get going with this system." In this study, we replaced "the system" with "Hipper" to capture the opinion of participants regarding the usability of our eHealth program
Oxford Hip Score (OHS) | Baseline, 7-10 days before surgery, Post Intervention (30 days after surgery)
  The OHS is a 12-item tool that assesses pain and function in patients undergoing hip replacement surgery. It demonstrates good construct validity and test-retest reliability in THR

CONTACTS AND LOCATIONS:
Overall Officials: William C Miller, PhD, Principal Investigator — University of British Columbia
Locations (1):
- GF Strong Rehabilitation Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohammadi S, Westby MD, Schneeberg A, Watson W, Dhariwal A, Simpson E, Miller WC. The hip instructional prehabilitation program for enhanced recovery (HIPPER) as an eHealth approach to presurgical hip replacement Education: Feasibility randomized controlled trial. Int J Orthop Trauma Nurs. 2025 Aug;58:101210. doi: 10.1016/j.ijotn.2025.101210. Epub 2025 Jun 18. PMID 40580786
- [Derived] Dhariwal A, Mohammadi S, Simpson E, Westby MD, Watson W, Miller WC. Patient-centered perspectives: A qualitative evaluation of the Hip Instructional Prehabilitation Program for Enhanced Recovery (HIPPER). PLoS One. 2025 Apr 24;20(4):e0322114. doi: 10.1371/journal.pone.0322114. eCollection 2025. PMID 40273090
- [Derived] Miller WC, Mohammadi S, Watson W, Crocker M, Westby M. The Hip Instructional Prehabilitation Program for Enhanced Recovery (HIPPER) as an eHealth Approach to Presurgical Hip Replacement Education: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Jul 6;10(7):e29322. doi: 10.2196/29322. PMID 34255722